CLINICAL TRIAL: NCT00243100
Title: A Phase 1 Study of Suberoylanilide Hydroxamic Acid (SAHA) in Combination With Gemcitabine in Patients With Epithelial Tumors
Brief Title: Vorinostat and Gemcitabine in Treating Patients With Metastatic or Unresectable Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00091; NCI-2009-00091 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000445401; 2005-0140 (Other: M D Anderson Cancer Center); 6865 (Other: CTEP); U01CA062461 (NIH)
Record Dates: First submitted 2005-10-20; First posted 2005-10-21 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Vorinostat; Gemcitabine

ARMS (1):
- Arm I (Experimental): Patients receive oral vorinostat (SAHA) once daily on days 1-14 and gemcitabine IV over 1-2 hours on days 3 and 10. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of SAHA and gemcitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. A minimum of 6 patients are treated at the MTD
  Interventions: Drug: vorinostat; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: vorinostat — Given orally
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar

SUMMARY:
This phase I trial is studying the side effects and best dose of vorinostat and gemcitabine in treating patients with metastatic or unresectable solid tumors. Drugs used in chemotherapy, such as vorinostat and gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Vorinostat may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the dose-limiting toxicity, maximum tolerated dose, and pharmacokinetics of vorinostat (SAHA) and gemcitabine in patients with metastatic or unresectable epithelial solid tumors.

SECONDARY OBJECTIVES:

II. Determine tumor activity of this regimen in these patients.

OUTLINE: This is a dose-escalation, open-label study.

Patients receive oral vorinostat (SAHA) once daily on days 1-14 and gemcitabine IV over 1-2 hours on days 3 and 10. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of SAHA and gemcitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. A minimum of 6 patients are treated at the MTD.

After completion of study treatment, patients are followed for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* ECOG 0-2 OR Karnofsky 60-100%
* AST and ALT =< 2.5 times ULN
* Bilirubin =< 1.5 times upper limit of normal (ULN)
* Platelet count >= 100,000/mm3
* Absolute neutrophil count >= 1,500/mm3
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Any number and type of prior chemotherapies are allowed including prior use of gemcitabine chemotherapy. A washout phase of at least 2 weeks since use of prior chemotherapy or radiation therapy, 6 weeks if the last regimen included nitrosoureas or mitomycin C, is required.
* Patients must have histologically confirmed epithelial malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
* Ability to understand and the willingness to sign a written informed consent document.
* Patients must have at least one measurable lesion as per the RECIST Criteria that can be accurately measured in at least one dimension, with minimum lesion size equal to or more than twice the slice thickness of the imaging study used.

Exclusion Criteria:

* No symptomatic congestive heart failure
* No cardiac arrhythmia
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No history of allergy, significant side effects, or poor tolerance to gemcitabine
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to vorinostat (SAHA)
* At least 2 weeks since prior radiotherapy
* Recovered from prior therapy
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other uncontrolled illness
* More than 2 weeks since prior valproic acid
* No other concurrent investigational drugs
* No other concurrent anticancer therapy
* Patients with known brain metastases are excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2005-11; Primary Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Maximally tolerated dose of a combination of SAHA and gemcitabine determined by dose-limiting toxicity as measured by NCI CTCAE v3.0 continuously | 21 days
Pharmacokinetics of SAHA | -0.5, 0.5, 1, 2, 2.5, 3, 4, 6 and 8 hours after day 1 dose; -0.5 hours day 2; and -0.5, 0.5, 1, 2, 2.5, 3, 4, 6 and 8 hours day 3

SECONDARY OUTCOMES:
Best overall response (complete + partial response rate) as measured radiologically by RECIST | Up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Gauri Varadhachary, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States